CLINICAL TRIAL: NCT00169377
Title: Study of the Effects of High Frequency Stimulation of the Subthalamic Stimulation in the Treatment of Severe Obsessive-compulsive Disorders
Brief Title: Subthalamic Nucleus (STN) Stimulation and Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marie-laure Welter (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor-Investigator, Marie-laure Welter, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P030422
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive compulsive disorder; deep brain stimulation; subthalamic nucleus
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Deep brain stimulation on followed by off
  Interventions: Procedure: deep brain stimulation; Procedure: No stimulation
- Group B (Sham Comparator): No stimulation, deep brain stimulation off followed by on
  Interventions: Procedure: deep brain stimulation; Procedure: No stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — Stimulator on followed by off
Procedure: No stimulation — Stimulator off followed by on

SUMMARY:
Obsessive-compulsive disorder is a disabling and frequent disorder. In some patients, the medical treatment is ineffective. The pathophysiology of this disease is still unknown. Some data suggest that basal ganglia dysfunction could participate in the occurrence of OCD. The aim of this study is to evaluate the efficacy of subthalamic nucleus high-frequency stimulation in patients with severe OCD.

ELIGIBILITY:
Inclusion Criteria:

* Severe obsessive-compulsive disorder

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Severe cognitive or behavioral disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Yale-Brown-Obession and Compulsion Scale (YBOCS) | 2 three-month periods
  YBOCS

SECONDARY OUTCOMES:
Global assessment of function (GAF) | 10 month follow-up but 2 3-month period for the cross-over
  GAF
Clinical Global Impression(CGI) | 10 month follow-up but 2 3-month period for the cross-over
  CGI
Montgomery and Asberg Depression Rating scale (MADRS) | 10 month follow-up but 2 3-month period for the cross-over
  MADRS
Hospital Anxiety Depression scale (HAD-S) | 10 month follow-up but 2 3-month period for the cross-over
  HAD-S
Sheehan Disability Scale (SDS) | 10 month follow-up but 2 3-month period for the cross-over
  SDS
Brief Scale for Anxiety (BABS) | 10 month follow-up but 2 3-month period for the cross-over
  BABS
Social Adjustment scale self-report (SAS-SR) | 10 month follow-up but 2 3-month period for the cross-over
  SAS-SR
neuropsychological tests | 10 month follow-up but 2 3-month period for the cross-over
  STROOP, apathy scales
adverse event | 10 month follow-up but 2 3-month period for the cross-over
  adverse event
Yale-Brown-Obession and Compulsion Scale (YBOCS) | observational follow-up at 22 month, 34 month and 46 month
Global assessment of function (GAF) | observational follow-up at 22 month, 34 month and 46 month
Clinical Global Impression(CGI) | observational follow-up at 22 month, 34 month and 46 month
Montgomery and Asberg Depression Rating scale (MADRS) | observational follow-up at 22 month, 34 month and 46 month
Hospital Anxiety Depression scale (HAD-S) | observational follow-up at 22 month, 34 month and 46 month
Sheehan Disability Scale (SDS) | observational follow-up at 22 month, 34 month and 46 month
Social Adjustment scale self-report (SAS-SR) | observational follow-up at 22 month, 34 month and 46 month
Quality of life (SF-36) | observational follow-up at 22 month, 34 month and 46 month
neuropsychological tests | observational follow-up at 22 month, 34 month and 46 month
adverse event | observational follow-up at 22 month, 34 month and 46 month
Stimulation parameters | observational follow-up at 22 month, 34 month and 46 month

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mallet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - Bordeaux
  - Clermont-Ferrand
  - Grenoble
  - Nantes
  - Nice
  - Centre d'Investigation Clinique-Hôpital Pitié-Salpêtrière, Paris
  - Saint-Anne, Paris
  - Poitiers
  - Rennes
  - Toulouse

REFERENCES:
- [Derived] Le Jeune F, Verin M, N'Diaye K, Drapier D, Leray E, Du Montcel ST, Baup N, Pelissolo A, Polosan M, Mallet L, Yelnik J, Devaux B, Fontaine D, Chereau I, Bourguignon A, Peron J, Sauleau P, Raoul S, Garin E, Krebs MO, Jaafari N, Millet B; French Stimulation dans le trouble obsessionnel compulsif (STOC) study group. Decrease of prefrontal metabolism after subthalamic stimulation in obsessive-compulsive disorder: a positron emission tomography study. Biol Psychiatry. 2010 Dec 1;68(11):1016-22. doi: 10.1016/j.biopsych.2010.06.033. Epub 2010 Oct 16. PMID 20951978
- [Derived] Bourredjem A, Pelissolo A, Rotge JY, Jaafari N, Machefaux S, Quentin S, Bui E, Bruno N, Pochon JB, Polosan M, Baup N, Papetti F, Chereau I, Arbus C, Mallet L, du Montcel ST; French "Stimulation dans le Trouble Obsessionnel Compulsif (STOC)" Study Group. A video Clinical Global Impression (CGI) in obsessive compulsive disorder. Psychiatry Res. 2011 Mar 30;186(1):117-22. doi: 10.1016/j.psychres.2010.06.021. Epub 2011 Feb 12. PMID 20621362
- [Derived] Mallet L, Polosan M, Jaafari N, Baup N, Welter ML, Fontaine D, du Montcel ST, Yelnik J, Chereau I, Arbus C, Raoul S, Aouizerate B, Damier P, Chabardes S, Czernecki V, Ardouin C, Krebs MO, Bardinet E, Chaynes P, Burbaud P, Cornu P, Derost P, Bougerol T, Bataille B, Mattei V, Dormont D, Devaux B, Verin M, Houeto JL, Pollak P, Benabid AL, Agid Y, Krack P, Millet B, Pelissolo A; STOC Study Group. Subthalamic nucleus stimulation in severe obsessive-compulsive disorder. N Engl J Med. 2008 Nov 13;359(20):2121-34. doi: 10.1056/NEJMoa0708514. PMID 19005196